CLINICAL TRIAL: NCT03451123
Title: FET-PET/MRI for Surgical Assessment of Pediatric Brain Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R17-077
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Pediatric Brain Tumors

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FET-PET/MRI (Experimental): O-(2-[F-18]FET)-L-tyrosine (FET) for brain PET/MRI
  Interventions: Drug: FET PET/MRI

INTERVENTIONS:
Drug: FET PET/MRI — FET PET/MRI scan before and after surgery

SUMMARY:
The primary objectives of this study are:

1. Determine the percentage of patients whose surgical plan would change with FET-PET/MRI compared to MRI alone.
2. Determine the percentage of patients who have residual tumor after surgery detected with FET-PET/MRI.

A secondary objective of this study is:

1) Perform preliminary correlations between the pre- and post-surgical metabolic tumor volumes measured with FET-PET/MRI to progression free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a known or suspected primary brain tumor with a non-enhancing component with planned standard of care surgical resection. Patients with newly diagnosed or recurrent brain tumors are eligible.
2. Tumors with non-enhancing regions will be defined as T2/FLAIR hyperintensity extending at least 0.5 cm beyond areas of enhancement as assessed by MRI.
3. Patient must be 18 years of age or younger at the time of study enrollment.
4. Patient must have measurable disease defined as tumor measurable in two perpendicular dimensions on MRI greater than 1 cm.
5. Patient must have a life expectancy greater than 8 weeks.
6. Patient must be able to undergo FET-PET/MRI without sedation.
7. Females with childbearing potential must have a negative urine β-hCG test on the day of procedure or a serum hCG test within 48 hours prior to the administration FET. Females who have not reached menarche will not require pregnancy testing.

Exclusion Criteria:

1. Patient must not be receiving an investigational or standard of care anti-cancer drug within 6 months prior to the FET-PET/MRI study.
2. Patient must not have received radiation therapy within the past 6 months.
3. Patient must not have a contraindication to contrast-enhanced MRI (e.g. renal insufficiency, incompatible implant).
4. Patient must not be pregnant or breast feeding.
5. Patient must not have been treated for another cancer within 5 years with the exception of cutaneous basal cell carcinoma or squamous cell carcinoma.
6. Patients must not have a history of brain metastases.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients whose surgical plan change with FET-PET/MRI compared to MRI alone. | 2 years
  Surgical planning will be performed prior to brain tumor resection based on MRI alone and then with FET-PET/MRI. The surgical margins will be compared and the percentage of patients whose surgical plans change with FET-PET/MRI will be calculated.
Percentage of patients who have residual tumor after surgery detected with FET-PET/MRI | 2 years
  The percentage of patients with residual tumor identified with FET-PET/MRI will be measured. This percentage will be compared to detection of residual tumor by MRI alone.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Advanced Imaging Facility, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No